CLINICAL TRIAL: NCT07100353
Title: Premature Infants' Developmental Function, Daily Living, Participation, and Quality of Life: A Longitudinal Study
Status: Active, not recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202201544B0
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Premature Infant
Keywords: Developmental Function; Daily Living; Participation; Quality of Life
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Samples with DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Full-term Children: This study will recruit 100 full-term children (ages 0-3) without neurological or developmental disorders for longitudinal follow-up.
- Premature Children: This study will recruit 350 pretmature children (born <37 weeks, ages 0-3) in stable treatment for longitudinal follow-up.

SUMMARY:
This study tracks the long-term development of premature infants to examine how birth profiles, risk factors, and physical functioning influence their activities, participation, and quality of life. It also identifies predictors of functional outcomes, evaluates assessment tool sensitivity, validates the General Movements Assessment (GMA) as a prognostic tool, and compares findings with the Taiwan Infant Development Database. The study hypothesizes that birth conditions and postnatal complications predict differences in development and well-being, that risk factors and physical function relate to participation and quality of life, and that the GMA will show reliable validity across disability categories.

ELIGIBILITY:
1. Premature Cases

Inclusion criteria:

1. Born before 37 weeks.
2. Aged 0-3 years.
3. Caregivers consent and agree to cooperate.
4. Stable condition with regular outpatient care, medication, and rehabilitation.

Exclusion criteria:

1. Acute illness (e.g., infection).
2. Parents/caregivers unable to communicate in Chinese.

2. Full-term Cases

Inclusion criteria:

1. Born at full term.
2. Aged 0-3 years.
3. No disease affecting neurophysiological development.
4. Caregivers consent and agree to cooperate.

Exclusion criteria:

1. Medical conditions affecting neurophysiological development (e.g., traumatic brain injury).
2. Neurodevelopmental disorders
3. Sensory perception disorders
4. Chromosomal abnormalities
5. Parents/caregivers unable to communicate in Chinese.

Ages: 0 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will recruit 100 full-term children and 350 premature children for a longitudinal follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Bayley scales of infant and Toddler Development- fourth edition, Bailey-IV | Baseline
Comprehensive Development Inventory for Infant and Toddlers (CDIIT) | Baseline
KIT Development and Health Questionnaire | Baseline
General Movements Assessment (GMA) | Baseline
PREMature Infant Index (PREMII) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan